CLINICAL TRIAL: NCT07115238
Title: A Phase 3, Multicenter Study to Evaluate the Efficacy and Safety of PET Visual Assessment Using XTR006 Injection for Detection of Brain Neurofibrillary Tangles (NFTs) in Elderly Subjects
Brief Title: Analysis of 18F-XTR006 PET Imaging in Cognitively Normal Subjects, and Patients With MCI and AD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STB-XTR006-301
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Neurofibrillary Tangle
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alzheimer's Disease (Experimental): AD subjects will undergo PET imaging using [18F]XTR006.
  Interventions: Drug: XTR006
- Mild Cognitive Impairment Due to Alzheimer's Disease (Experimental): MCI subjects will undergo PET imaging using [18F]XTR006.
  Interventions: Drug: XTR006
- Cognitively normal (Experimental): Cognitively normal subjects will undergo PET imaging using [18F]XTR006.
  Interventions: Drug: XTR006

INTERVENTIONS:
Drug: XTR006 — all patients will receive one injection of [18F]XTR006, a PET radiopharmaceutical selective for NFTs. For the injection, subjects will receive a target dose of 4-6 mCi IV as a bolus injection. [18F]XTR006 injection will be followed by a 10 ml saline flush.
  Other Names: [18F]MK 6240; Florquinitau

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of XTR006 injection PET visual reading in detecting brain neurofibrillary tangles (NFTs) in elderly subjects with Mild Cognitive Impairment (MCI), Alzheimer's Disease (AD), and cognitively normal individuals. The main question it aims to answer is:

• What is the sensitivity and specificity of XTR006 PET visual reading results compared to the truth standard across MCI, AD, and cognitively normal subjects?

Participants will:

* Receive XTR006 injection
* Undergo PET/CT scanning

DETAILED DESCRIPTION:
This is a multicenter, single-blind, non-randomized phase III study. The study aims to evaluate the effectiveness of XTR006 PET imaging visual reads for detecting NFTs in subjects. The trial procedures for all subjects include a screening period, an administration period, and a follow-up period. All subjects must sign an informed consent form before entering the screening period.

In this study, nuclear medicine physicians with tau-PET image reading experience will undergo training in the XTR006 PET visual reading methodology. Three nuclear medicine physicians who achieve excellent scores on the assessment will be selected as blinded visual readers for this study. All subject images will be visually interpreted in a blinded manner according to the XTR006 PET visual reading methodology. The final reading conclusion will be determined by consensus of at least two blinded visual readers. Using the composite diagnostic results of clinical cognitive assessment and Aβ-PET examination as the reference standard, sensitivity and specificity will be calculated with their 95% confidence intervals. The primary endpoint of this study will be considered achieved if the lower limit of the confidence interval exceeds the target value of 60%. Additionally, this study will analyze PET SUVR across groups to evaluate XTR006 uptake characteristics in different populations from a semi-quantitative perspective and assess the safety of XTR006 through analysis of post-administration AEs and SAEs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Subjects:

1. Male or female subjects aged ≥50 years.
2. Able to tolerate both PET and MRI examinations.
3. Must use contraceptive measures during the study period and for 6 months after study completion.
4. Written informed consent must be obtained before any assessment is performed.

Inclusion Criteria for Cognitively Normal Subjects:

1)CDR (Clinical Dementia Rating) score of 0. 2）MMSE (Mini-Mental State Examination) score ≥28. 3）Negative visual reading result on brain Aβ-PET imaging.

Inclusion Criteria for Subjects with MCI:

1. Meet the core clinical criteria for MCI due to AD according to 2011 NIA-AA (National Institute on Aging-Alzheimer's Association) standards
2. Positive visual reading result on brain Aβ-PET imaging

Inclusion Criteria for Subjects with AD:

1. Meet the specific clinical phenotype criteria for typical AD according to 2014 International Working Group (IWG)-2 standards:
2. Positive visual reading result on brain Aβ-PET imaging.

Exclusion Criteria:

1. Diagnosis of atypical AD, frontotemporal lobar degeneration (FTLD), Lewy body dementia, or other types of dementia.
2. Current significant psychiatric illness with symptoms that prevent completion of imaging procedures.
3. MRI-confirmed structural brain abnormalities, such as large stroke or intracranial mass lesions.
4. Claustrophobia.
5. History of alcohol abuse or drug abuse/dependence.
6. Allergy to the study drug or any of its components.
7. Women who are currently breastfeeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of visual reading of XTR006 PET imaging in detecting tau NFTs (neurofibrillary tangles) | 12month
  The sensitivity and specificity of XTR006 PET imaging visual reading results compared to the truth standard.

SECONDARY OUTCOMES:
Compare the overall brain uptake patterns of XTR006 in MCI (Mild Cognitive Impairment), AD (Alzheimer's Disease), and cognitively normal subjects. | 12month
  The inter-group differences in XTR006 PET Standardized Uptake Value Ratios (SUVR) within brain regions of interest(ROIs) among different subject groups；The sensitivity and specificity of semi-quantitative SUVR analysis in differentiating between different subject groups.
Safety and Tolerability Profile Measured by Adverse Events (AEs) | 12month
  Safety and tolerability profile for the administration of [18F]XTR006 and PET scanning are measured by number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Shi, Doctor, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided